CLINICAL TRIAL: NCT02869217
Title: Phase Ib Study of TBI-1301 (NY-ESO-1 Specific TCR Gene Transduced Autologous T Lymphocytes) in Patients With Solid Tumors
Brief Title: Study of TBI-1301 (NY-ESO-1 Specific TCR Gene Transduced Autologous T Lymphocytes) in Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1301-02
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: NY-ESO-1 Expressing Solid Tumors in HLA-A2 Positive Patients; Synovial Sarcoma; Melanoma; Esophageal Cancer; Ovarian Cancer; Lung Cancer; Bladder Cancer; Liver Cancer
Keywords: NY-ESO-1 expressing solid tumors in HLA-A2 positive patients
MeSH Terms: conditions — Sarcoma, Synovial; Melanoma; Esophageal Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Liver Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort B (retreatment) (Experimental): Cyclophosphamide will be given intravenously (by vein) at a fixed dose of 750mg/m^2/d for 2 days.
  Fludarabine will be given intravenously at a fixed dose of 30mg/m^2/d for 2 days.
  TBI-1301 cells will be infused on Day 0 at a dose of 5x10^9 cells.
  *Patients will only enter into this cohort if they have already been enrolled in another cohort prior
  Interventions: Drug: Cyclophosphamide; Biological: TBI-1301; Drug: Fludarabine
- Cohort C (double infusion) (Experimental): Cyclophosphamide will be given intravenously (by vein) at a fixed dose of 750mg/m^2/d for 2 days.
  Fludarabine will be given intravenously at a fixed dose of 30mg/m^2/d for 2 days.
  TBI-1301 cells will be infused on Day 0 and Day 14 at a dose of 5x10^9 cells.
  Interventions: Drug: Cyclophosphamide; Biological: TBI-1301; Drug: Fludarabine

INTERVENTIONS:
Drug: Cyclophosphamide
Biological: TBI-1301
Drug: Fludarabine

SUMMARY:
The target populations for this phase I study with TBI-1301 are patients with advanced solid tumors. Patients' tumors will be required to express NY-ESO-1, which include but is not limited to ovarian cancer, synovial sarcoma, esophageal cancer, lung cancer, bladder cancer, liver cancer, and malignant melanoma. Patients must be positive for HLA-A*02:01 or HLA-A*02:06 and the patient's tumor tissue must be positive for NY-ESO-1 antigen expression. The study will take the subject's T cells, which are a natural type of immune cell in the blood, and send them to a laboratory to be modified. The changed T cells used in this study will be the subject's own T cells that have been genetically changed with the aim of attacking and destroying cancer cells.

The manufacturing of T cells takes about 1 month to complete. The T cells will be given back to the subject through an intravenous infusion. The purpose of this study is to test the safety of genetically changed T cells and find out what effects, if any, they have in subjects with advanced solid tumors.

The purpose of this study is to evaluate the safety profile of TBI-1301, to determine the recommended phase 2 (RP2D) dose of TBI-1301 when administered following cyclophosphamide and fludarabine pre-treatment, to evaluate the safety of repeat dosing of TBI-1301, to assess the presence/absence of RCR appearance after TBI-1301 infusion, to assess the presence or absence of clonality by LAM-PCR, and to evaluate evidence of efficacy of TBI-1301 using RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or recurrent unresectable solid tumor.
* HLA-A*02:01 or HLA-A*02:06 positive.
* Tumor NY-ESO-1 expression by immunohistochemistry.
* No anti-cancer chemotherapy, radiation therapy or immunotherapy within 2 weeks or 5 half-lives of PBMC harvest.
* The treating investigator should consider the patient to have disease that is incurable and that the patient would be a reasonable candidate for future treatment with TBI-1301.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >10 mm with CT scan, MRI, or calipers by clinical exam. Patients must have radiographic evidence of disease progression following the most recent line of treatment. Areas of previous radiation may not serve as measurable disease unless there is evidence of progression post radiation.
* ECOG Performance Status 0 or 1.
* Age ≥16 years on consent.
* Life expectancy greater than 4 months.
* The following laboratory requirements must be met (within 14 days prior to phlebotomy for generation of TBI-1301):
* Absolute neutrophil count (ANC) ≥1.5 x10^9/L (1500/μL) without G-CSF support
* WBC ≥ 2.5x10^9/L (2,500/μl)
* Lymphocytes ≥ 0.5x10^9/L (500/μl)
* Hemoglobin ≥ 80 g/L
* Platelets ≥ 75x10^9/L (75,000/μl)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (≤2.5X if Gilbert's disease)
* AST(SGOT), ALT(SGPT) < 3.0 x ULN (< 5 x ULN with known liver metastases)
* Creatinine ≥ 60 ml/min (calculated by Cockcroft and Gault)
* Adequate renal function
* Consent must be appropriately obtained in accordance with applicable local and regulatory requirements.

Exclusion Criteria:

* Uncontrolled intercurrent illnesses or medical conditions that may interfere with trial participation such as ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, severe active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement or compromise the ability of the subject to give written informed consent.
* Patients who are receiving any other investigational agents.
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Subjects with vitiligo, Grave's disease, Hashimoto's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
* No evidence of active uncontrolled infection (patients on antibiotics are eligible).
* History of primary immunodeficiency.
* History of organ transplant that requires use of immunosuppressives.
* Known allergy or reaction to a known component of TBI-1301.
* Untreated central nervous system metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and/or corticosteroids. If treated lesions are shown to be stable for 1 month the subject may be eligible.
* Other invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured.
* Current or prior use of immunosuppressive medication within 14 days before phlebotomy, with the exceptions of intranasal, topical, and inhaled corticosteroids or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent. Oral steroid use as premedication to prevent allergic reactions to radiologic contrast is allowed.
* Any condition that, in the opinion of the investigator, would interfere with the evaluation of TBI-1301 or interpretation of subject safety or study results.
* Known history of tuberculosis.
* HIV positive.
* Active HTLV or syphilis infection.
* Active hepatitis B infection (hepatitis B surface antigen or HBV DNA positive).
* Active hepatitis C infection (if hepatitis C antibody positive, HCV RNA positive).
* Has no known active central nervous system metastases and/or carcinomatous meningitis.
* Ongoing prior toxicities related to previous anti-cancer treatments (surgery, radiotherapy or adjuvant chemo-radiation) must be recovered to < grade 1 or baseline
* Pregnant women are excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-09; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Safety profile (i.e. adverse events, presence/absence of RCR, analysis of clonality and PK of TBI-1301) assessed by CTCAE v.4.0 and laboratory testings. | 8 weeks
Recommended phase 2 (RP2D) dose o TBI-1301 when administered following cyclophosphamide and fludarabine pre-treatment | 8 weeks

SECONDARY OUTCOMES:
Evidence of efficacy (i.e. anti-tumor effect) of TBI-1301 measured using RECIST v1.1 | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada